## THE IMPACT OF INTRAOPERATIVE LIDOCAINE INFUSION ON POSTOPERATIVE RECOVERY AFTER HYSTEROSCOPY: A RANDOMIZED CONTROLLED TRIAL

## INFORMED CONSENT FORM 26th FEBRUARY 2024

## INFORMED VOLUNTARY CONSENT FORM

The study you are participating in is a scientific research and the name of the research is "The effectiveness of intravenous lidocaine treatment in post-operative pain control in patients undergoing hysteroscopy."

Hysteroscopy is a frequently used method in the diagnosis and treatment of pathologies such as abnormal uterine bleeding, infertility, endometrial pathologies, uterine fibroids, and intrauterine synechia. General Anesthesia (GA) is the frequently preferred method in operative hysteroscopy. Intraoperative lidocaine infusion is a frequently preferred method in surgical procedures because it reduces the need for opioids, provides better postoperative pain control, reduces postoperative nausea and vomiting, and increases rapid recovery. This method has been shown to reduce complications such as postoperative pain after procedures such as endoscopic submucosal dissection and laparoscopic cholecystectomy. Our aim in this study is to show the effect of intraoperative lidocaine infusion in reducing complications such as pain, nausea, vomiting, and opioid analgesia requirement after hysteroscopy operations frequently performed in gynecology clinics. Participation in this study is entirely voluntary. You may decline to participate in the study; this situation will not lead to any penalty or hindrance to your benefits. The results of the research will be used for scientific purposes. Medical data about you may also be used for scientific purposes if necessary.

You can leave the study at any time. Your information will not be shared with anyone in any way. You can reach the doctors involved in the study from our hospital's phone number 05467240341.

All your medical and identity information will be kept confidential and your identity information will not be given even if the study is published, but the audience of the study, those conducting the examination, ethics committees and official authorities can access your medical information when necessary. You can also access your own medical information whenever you want.

## **Consent to Participate in the Study:**

I have read and listened to the information provided above, which should be given to the volunteer before starting the research. I have asked the researcher all the questions that come to my mind, and I have understood in detail all the explanations given to me in written and verbal form. I have been given sufficient time to decide whether I want to participate in the study. Under these conditions, I authorize the researcher to review, transfer and process my medical information, and I accept the invitation to participate in the study voluntarily, without any coercion or pressure.

A signed copy of this form will be given to me.